CLINICAL TRIAL: NCT04176601
Title: Engage Psychotherapy to Promote Connectedness in Caregivers: A Pilot Study of the Rochester Roybal Center for Social Ties and Aging Research
Brief Title: Engage Psychotherapy to Promote Connectedness in Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kimberly Van Orden, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P30AG064103-Pilot2; P30AG064103 (NIH)
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Loneliness; Social Isolation; Caregiver Burnout
MeSH Terms: conditions — Social Isolation; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engage Coaching (Experimental): Engage Coaching helps caregivers bolster motivation for increasing connectedness, teaches problem solving skills, and provides behavioral practice with social engagement. Up to 8 brief sessions (typically 30 minutes) are provided weekly over no more than three months.
  Interventions: Behavioral: Engage coaching

INTERVENTIONS:
Behavioral: Engage coaching — Participants will complete up to 8 weekly individual Social Engage psychotherapy sessions. Participants will be allotted up to 3 months to complete all sessions, a time-frame that allows for two weeks without meeting to address life stressors such as illnesses that may pop up. All sessions are provided via phone or videocall (Zoom). The first and last session are longer - up to 60 minutes if needed. Middle sessions are shorter (20-45 minutes). Engage is a stepped care psychotherapy in that the simplest strategy is taught first-action planning (a derivative of problem solving therapy)-and "barrier strategies" are added only if needed. Action plans are designed to address loneliness and social isolation in the context of caregiving demands.

SUMMARY:
The Engage Coaching Project is a Stage 1 intervention development study. This study asks: "what behavioral strategies are needed to help socially disconnected caregivers with significant barriers to increasing connectedness?" This study uses a mixed methods approach to adapt a brief behavioral intervention-Social Engage psychotherapy-for use with socially disconnected caregivers. The ultimate goal is for Social Engage psychotherapy to be offered as a second step in a stepped care approach for caregivers who do not demonstrate an adequate response to a single-session psychoeducation plus resources intervention. Social Engage Psychotherapy helps caregivers bolster motivation for increasing connectedness, teaches problem solving skills, and provides behavioral practice with social engagement. Up to 8 brief sessions (typically 30 minutes) are provided weekly over no more than three months. This is a single-arm clinical trial of Social Engage psychotherapy, with up to 30 participants.

DETAILED DESCRIPTION:
This is a Stage 1 intervention development study. This study asks: "what behavioral strategies are needed to help socially disconnected caregivers with significant barriers to increasing connectedness?" Pilot 2 uses a mixed methods approach to adapt a brief behavioral intervention-Social Engage psychotherapy-for use with socially disconnected caregivers, which we call Engage Coaching for Caregivers. The ultimate goal is for Engage Coaching for Caregivers to be offered as a second step in a stepped care approach for caregivers who do not demonstrate an adequate response to a single-session psychoeducation plus resources intervention. Engage Coaching helps caregivers bolster motivation for increasing connectedness, teaches problem solving skills, and provides behavioral practice with social engagement. Up to 8 brief sessions (typically 30 minutes) are provided weekly over no more than three months. This is a single-arm clinical trial with up to 30 participants. The study's primary objective is to discover the most useful strategies to promote social connectedness in the context of caregiving. Participants will complete up to 8 weekly individual Engage Coaching sessions via phone or Zoom. Participants will be allotted up to 3 months to complete all sessions, a time-frame that allows for two weeks without meeting to address life stressors such as illnesses that may pop up. The first and last session are longer - up to 60 minutes if needed. Middle sessions are shorter (20-45 minutes). Engage is a stepped care psychotherapy in that the simplest strategy is taught first-action planning (a derivative of problem solving therapy)-and "barrier strategies" are added only if needed. Coaches and the PI will work together to devise caregiver specific barrier strategies as needed, such as brief communication skills coaching or education on behavioral issues in dementia. The development and piloting of these new caregiver specific barrier strategies is a key objective of this pilot study. During the data analysis phase, we will conduct qualitative analyses from participants on which of these strategies were most useful and combined with experiences from therapists, we will adapt the therapy manual to include the most useful strategies, for testing in a subsequent Stage II efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 yrs;
2. English speaking;
3. Caregiver for a community-dwelling family member with ADRD, living with (or in close proximity to) family member with dementia;
4. Endorse elevated caregiving distress as measured by a score of greater than 11 on the 10-item Perceived Stress Scale (PSS-10) and/or a score of 5 or greater on the Modified Caregiver Strain Index (MCSI);
5. Endorse clinically significant loneliness as measured by a score of greater than 6 on the UCLA Loneliness Scale: Short Form.

Exclusion Criteria:

1. Primary language is not English;
2. Recent or current psychosis;
3. Significant cognitive impairment;
4. Hearing problems that preclude completion of the intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Van Orden, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic and health history data from interviews with 30 older adults who are caregivers for individuals with ADRD and transcribed responses to semi-structured interviews. Data from this research will be made available to the public in the University of Rochester's institutional repository, UR Research, at https://urresearch.rochester.edu. We will share the research protocols, in a text format, such as MS Word or PDF. Qualitative data will also be made available in text form. For quantitative data, the PI will make available the actual datasets generated from research, in a commonly- used format such as a SAS® dataset. The datasets will be associated with a related publication, research protocol or other documentation of the original research. Some research data may be in multimedia form (such as recordings of focus group sessions).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Timetable to release the data: the data and referenced resources from publications will be made available by the on-line publication date.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement as suggested by the NIH that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. 4. De-identification of data from human subjects: A final complete database will be created to host all data which will be stripped of any identifiers and stored pursuant to UR Institutional Review Board protocols. Confidentiality for research subjects for qualitative data will be promoted by the use of an anonymization scheme and anonymizing the data as the qualitative files are created for the analysis (following guidelines developed by the Inter-university Consortium for Political and Social Research, 2012).
URL: https://urresearch.rochester.edu

REFERENCES:
- [Result] Van Orden KA, Bower E, Lutz J, Silva C. Engage coaching for caregivers: a pilot trial to reduce loneliness in dementia caregivers. Aging Ment Health. 2023 Sep-Oct;27(10):2019-2026. doi: 10.1080/13607863.2023.2187345. Epub 2023 Mar 10. PMID 36898849

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engage Coaching
Started | 30
Completed | 25
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Engage Coaching
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.37 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Loneliness
Description: UCLA Loneliness Scale Version 3, which assesses self-reported loneliness. 20 items, rated as to how often the participant has felt a certain way in the prior month (e.g., "How often do you feel alone?") -- "never" (1), "rarely" (2), "sometimes" (3), or "often" (4). Higher scores indicate greater loneliness. However, some individual items must be reverse-coded so that higher total scores reflect greater loneliness (i.e., 1=4, 2=3, 3=2, 4=1). These items (e.g., "How often do you feel there are people you can turn to?") are items 1,5,6,9,10,15,16,19,20. Total scores range from 20 to 80, with higher scores representing a worse outcome (i.e., greater loneliness).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage Coaching
Number analyzed (Participants) | 25
units on a scale
  Loneliness at baseline | 48.76 (10.04)
  Loneliness at 3 months | 44.44 (10.01)
Statistical Analysis 1: Comparison: Engage Coaching; Test type: Superiority; Mean Difference (Net) = 4.32, 95% CI 2-sided [1.49 to 7.15], Standard Error of Mean 1.37

2. Primary Outcome: Social Functioning
Description: Satisfaction with Social Roles and Activities (PROMIS) is a computerized adaptive test (CAT). It produces T scores with a mean of 50 and standard deviation of 10. Greater scores indicate better outcomes (i.e., greater satisfaction with social role and activities).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage Coaching
Number analyzed (Participants) | 25
units on a scale
  Social functioning at baseline | 40.22 (5.25)
  Social functioning at 3 months | 44.92 (6.75)
Statistical Analysis 1: Comparison: Engage Coaching; Test type: Superiority; Mean Difference (Net) = 4.70, 95% CI 2-sided [1.26 to 8.15], Standard Error of Mean 1.67

3. Secondary Outcome: Perceived Social Isolation
Description: PROMIS Perceived Social Isolation Computerized Adaptive Test. This is a computerized adaptive test (CAT) that assessed perceived social isolation. It produces T scores with a mean of 50 and standard deviation of 10. Greater scores indicate worse outcomes (i.e., greater perceived social isolation).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage Coaching
Number analyzed (Participants) | 25
score on a scale
  Perceived social isolation baseline | 54.61 (6.21)
  Perceived social isolation 3 months | 50.74 (6.01)
Statistical Analysis 1: Comparison: Engage Coaching; Test type: Superiority; Mean Difference (Net) = 3.68, 95% CI 2-sided [1.59 to 6.14], Standard Error of Mean 1.10

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Engage Coaching
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT04176601/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT04176601/SAP_001.pdf